CLINICAL TRIAL: NCT03820388
Title: Comparison of Etomidate Plus Propofol, Etomidate Alone on Induction of Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 909765
Record Dates: First submitted 2018-01-09; First posted 2019-01-29 (Actual); Results first posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Surgery
Keywords: Etomidate; Propofol
MeSH Terms: interventions — Propofol; Etomidate

STUDY DESIGN:
Intervention Model Description: Patients in 3 cohorts will be administered 30 second bolus by manual hand push
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Propofol Group (Experimental): Propofol 2 mg/kg
  Interventions: Drug: Propofol 2mg/kg
- Etomidate Group (Experimental): Etomidate 0.3 mg/kg
  Interventions: Drug: Etomidate 0.3 mg/kg
- Propofol plus Etomidate Group (Experimental): Propofol 1 mg/kg plus Etomidate 0.15 mg/kg
  Interventions: Drug: Propofol 1 mg/kg; Drug: Etomidate 0.15 mg/kg

INTERVENTIONS:
Drug: Propofol 2mg/kg — 2 mg/kg
  Other Names: Diprivan
  Arms: Propofol Group
Drug: Etomidate 0.3 mg/kg — 0.3 mg/kg
  Other Names: Amidate
  Arms: Etomidate Group
Drug: Propofol 1 mg/kg — 1 mg/kg Propofol
  Other Names: Diprivan
  Arms: Propofol plus Etomidate Group
Drug: Etomidate 0.15 mg/kg — 0.15 mg/kg Etomidate
  Other Names: Amidate
  Arms: Propofol plus Etomidate Group

SUMMARY:
Comparison of Etomidate plus Propofol vs. Propofol or Etomidate alone during induction of anesthesia.

DETAILED DESCRIPTION:
Comparison of Etomidate plus Propofol vs. Propofol or Etomidate alone during induction of anesthesia. The specific aims are testing patient reactions during induction, and in the post-anesthesia care unit (PACU).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective non-cardiac surgery
* ASA physical status of 2 or 3
* Age equal to or greater than 18 years old

Exclusion Criteria:

* Adults unable to provide consent
* Age less than 18 years old
* Pregnant women
* Prisoners
* Difficult airway
* Morbid Obesity
* Preoperative sedation use
* Severe Cardiac, pulmonary and liver disease
* Hypotension and shock
* Emergency surgeries
* Allergy to propofol or etomidate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2018-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hong Liu, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Propofol Group | Etomidate Group | Propofol Plus Etomidate Group
Started | 25 | 25 | 25
Completed | 25 | 25 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propofol Group | Etomidate Group | Propofol Plus Etomidate Group | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (8.5) | 62.5 (14.7) | 61.4 (11.6) | 61.7 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 12 | 39
  Male | 11 | 12 | 13 | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 25 | 75

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure
Description: Blood Pressure Fluctuations during Induction; change of blood pressure from baseline from induction to 10 min after induction.
Time Frame: 10 minutes after induction (intraoperative)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Propofol Group | Etomidate Group | Propofol Plus Etomidate Group
Number analyzed (Participants) | 25 | 25 | 25
mmHg | 105 (16) | 122 (23) | 117.88 (18)

2. Primary Outcome: Heart Rate
Description: Heart Rate changes during induction (Beats Per min)
Time Frame: 10 minutes after induction (intraoperative)
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Propofol Group | Etomidate Group | Propofol Plus Etomidate Group
Number analyzed (Participants) | 25 | 25 | 25
bpm | 77 (17) | 74 (12) | 74 (11)

3. Secondary Outcome: Pain at Injection Site
Description: Pain on injection will be measured using 4 graded scale; 0 = no pain, 1 = verbal complaint of pain, 2 = withdrawal of arm, 3 = both verbal complaint and withdrawal of arm.
Time Frame: intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Propofol Group | Etomidate Group | Propofol Plus Etomidate Group
Number analyzed (Participants) | 25 | 25 | 25
Participants | 7 | 0 | 0

4. Secondary Outcome: Myoclonic Movements
Description: The incidence and degree of myoclonic movements also recorded as follows: 0 = no myoclonic movements, 1 = minor myoclonic movements, 2 = moderate myoclonic movements, 3 = major myoclonic movements.
Time Frame: intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Propofol Group | Etomidate Group | Propofol Plus Etomidate Group
Number analyzed (Participants) | 25 | 25 | 25
Participants | 1 | 6 | 1

5. Secondary Outcome: Post-operative Nausea and Vomiting
Description: Presence of post-operative nausea or vomiting (yes/no).
Time Frame: 24 hours post-operation
Measure: Count of Participants; unit: Participants
Arm/Group | Propofol Group | Etomidate Group | Propofol Plus Etomidate Group
Number analyzed (Participants) | 25 | 25 | 25
Participants | 0 | 1 | 2

6. Secondary Outcome: Sedation Depth
Description: Sedation depth using bispectral index (BIS). BIS scores range from 0-100. A value of 0 indicates no EEG activity, 40-60 indicates an appropriate level of general anesthesia, and 90-100 is typical of a state of wakefulness.
Time Frame: 30 minutes post-induction
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Propofol Group | Etomidate Group | Propofol Plus Etomidate Group
Number analyzed (Participants) | 25 | 25 | 25
units on a scale | 30 (8.4) | 38 (11) | 38 (13)

7. Secondary Outcome: Eyelash Reflex Disappear Time
Description: Time to disappearance of eyelash reflex after induction.
Time Frame: Post induction, up to 1 hour
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Propofol Group | Etomidate Group | Propofol Plus Etomidate Group
Number analyzed (Participants) | 25 | 25 | 25
minutes | 31.9 (8.3) | 34.5 (7.5) | 32.4 (9)

8. Secondary Outcome: Intubation Time
Description: Duration of orotracheal intubation.
Time Frame: Up to 2 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Propofol Group | Etomidate Group | Propofol Plus Etomidate Group
Number analyzed (Participants) | 25 | 25 | 25
minutes | 92 (9.6) | 95 (8.9) | 93 (9.5)

ADVERSE EVENTS:
Time Frame: duration in-hospital up to 24 hours
Arm/Group | Propofol Group | Etomidate Group | Propofol Plus Etomidate Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT03820388/Prot_003.pdf
  • Statistical Analysis Plan (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/88/NCT03820388/SAP_004.pdf
  • Informed Consent Form (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/88/NCT03820388/ICF_005.pdf